CLINICAL TRIAL: NCT06409897
Title: Respiratory Mechanics Assessment at Different Head of the Bed Elevations in Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 68464523.9.0000.0068
Record Dates: First submitted 2024-04-24; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Failure; Pulmonary Disease
Keywords: Respiratory Failure; Pulmonary disease; Intensive care; Respiratory Mechanics
MeSH Terms: conditions — Respiratory Insufficiency; Lung Diseases

STUDY DESIGN:
Intervention Model Description: All the participants will be exposed to the same situations (head-of-bed elevations), in the same order. An alveolar recruitment maneuver followed by a PEEP titration with 10-degree head-of-bed elevation will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential head-of-bed elevation (Other): Patients will be positioned at 0 degrees of head-of-bed elevation, and after stabilization of the plethysmogram, data from electrical impedance tomography, hemodynamics, and arterial blood gas will be collected (arterial blood will be drawn by a nurse or physician). Sequentially and in the same manner, the bed will be adjusted to 10, 20, 30, and 40 degrees (the same data will be collected, except for the arterial blood sample, which will only be collected at the 40-degree elevation). Then, an alveolar recruitment maneuver will be performed, followed by a PEEP titration with 10-degree of head-of-bed elevation, and the data will be collected just as in the 0° and 40° steps.
  Interventions: Other: Sequencial increasing of head of the bed elevation and alveolar recruitment maneuver followed by a PEEP titration with 10° of head of the elevation

INTERVENTIONS:
Other: Sequencial increasing of head of the bed elevation and alveolar recruitment maneuver followed by a PEEP titration with 10° of head of the elevation — Patients will be sequentially positioned at 0, 10, 20, 30, and 40 degrees of head-of-bed elevation. An alveolar recruitment maneuver will be performed. For patients with body mass index ≤ 30 kg/m^2, the maneuver will be conducted in pressure control mode, pressure control = 15 cmH2O, respiratory rate = 20 breaths per minute, and the PEEP will be increased in steps of 5 up to 30 cmH2O. For patients with body mass index > 30, the PEEP will be increased up to 35. Then, a PEEP titration will be performed, tidal volume = 5 mL/Kg, respiratory rate = 25 breaths per minute, and the PEEP will be decreased from 24 down to 4 cmH2O in steps of 2 cmH2O with 30 seconds in each PEEP level. The PEEP titration software of Enlight 2100 will be used to determine the ideal PEEP, defined as the PEEP level with a collapse less than 5%. The alveolar recruitment maneuver will be performed again to reopen the lungs. Then, data will be collected, as with the 0 and 40-degree steps, with ideal PEEP.

SUMMARY:
The effects of different degrees of head-of-bed elevation on respiratory mechanics are poorly explored in the literature, and no study has investigated such effects using electrical impedance tomography, esophageal and gastric balloons to identify the ideal angle for optimizing respiratory mechanics. The hypothesis is that there is a optimal degree for the respiratory mechanics.

DETAILED DESCRIPTION:
Respiratory mechanics and regional ventilation will be monitored using electrical impedance tomography (Enlight 2100, Timpel Medical®, Brazil) . Esophageal and gastric pressures will be obtained through esophageal and gastric balloon catheters (Nutrivent®) (validation concerning to modified Baydur maneuver - slope delta esophageal pressure/delta airway pressure (0,8-1,2). We are using the hardware Pneumodrive (Biônica, Recife, Brazil) to record and store the esophageal, gastric and airway pressures, these data will be analyzed using LabVIEW 7.1 (Pneumobench).

Initially, patients will be positioned at 0 degrees of head-of-bed elevation, and after stabilization of the plethysmogram, data from electrical impedance tomography, hemodynamics, and arterial blood gas will be collected (arterial blood will be drawn by a nurse or physician). Sequentially and in the same manner, the bed will be adjusted to 10, 20, 30, and 40 degrees (the same data will be collected, except for the arterial blood sample, which will only be collected at the 40-degree elevation). Then, an alveolar recruitment maneuver will be performed, followed by a PEEP titration with 10-degree of head-of-bed elevation.

ELIGIBILITY:
Inclusion Criteria:

* Patients under invasive mechanical ventilation, intubated due to respiratory failure

Exclusion Criteria:

* Hemodynamics instability, contraindication for monitoring with esophageal and gastric catheters, and Electrical impedance tomography, no authorization of medical team of the intensive care unit, and contraindication for lung recruitment maneuver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory system compliance | At 0, 10, 20, 30, 40-degrees of head-of-bed elevation, and with titrated PEEP at 10-degrees of head-of-bed elevation
  Respiratory system compliance (mL/cmH2O) will be measured using electrical impedance tomography monitoring (Enlight 2100, Timpel Medical®, Brazil).
Lung compliance | At 0, 10, 20, 30, 40-degrees of head-of-bed elevation, and with titrated PEEP at 10-degrees of head-of-bed elevation
  Lung compliance (mL/cmH2O) will be measured offline using the esophageal pressure tracings. By knowing the respiratory system and chest wall compliance, the lung compliance will be calculated. (1/respiratory system compliance = 1/chest wall compliance + 1/lung compliance)
Chest wall compliance | At 0, 10, 20, 30, 40-degrees of head-of-bed elevation, and with titrated PEEP at 10-degrees of head-of-bed elevation
  Chest wall compliance (mL/cmH2O) will be measured offline using the esophageal pressure tracings.
  Chest wall compliance = tidal volume / delta esophageal pressure

SECONDARY OUTCOMES:
Oxygenation | At 0 and 40-degrees of head-of-bed elevation, and with titrated PEEP at 10-degrees of head-of-bed elevation
  Oxigenation will be assessed using the partial pressure arterial oxygen/fraction inspired oxygen ratio. Partial pressure arterial oxygen measured in the blood sample at the of each step and the fraction inspired oxygen set during the blood sample collection will be used.
Pressure between patient skin surface and the mattress | At 0, 10, 20, 30, 40-degrees of head-of-bed elevation
  ForeSite PT (XSENSOR Technology Corporation, Patient Monitoring System) will be used to measure the pressure between patient's skin surface and the mattress. A monitor connected to this sensor provides continuous pressure monitoring, and the data will exported for subsequent offline analysis of the sacral and occipital regions.
Hemodynamics satefy of keeping low degrees of head of the elevation | At 0, 10, 20, 30, 40-degrees of head-of-bed elevation
  Arterial blood pressure provided by the multiparameter monitor. Data will be noted in each degree.
Gastric pressure | At 0 and 40-degrees of head-of-bed elevation, and with titrated PEEP at 10-degrees of head-of-bed elevation
  Gastric pressure will be measured offline using the gastric pressure tracings.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo BP Amato, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Villar J, Kacmarek RM, Perez-Mendez L, Aguirre-Jaime A. A high positive end-expiratory pressure, low tidal volume ventilatory strategy improves outcome in persistent acute respiratory distress syndrome: a randomized, controlled trial. Crit Care Med. 2006 May;34(5):1311-8. doi: 10.1097/01.CCM.0000215598.84885.01. PMID 16557151
- [Background] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Costa EL, Lima RG, Amato MB. Electrical impedance tomography. Curr Opin Crit Care. 2009 Feb;15(1):18-24. doi: 10.1097/mcc.0b013e3283220e8c. PMID 19186406
- [Background] Galiatsou E, Kostanti E, Svarna E, Kitsakos A, Koulouras V, Efremidis SC, Nakos G. Prone position augments recruitment and prevents alveolar overinflation in acute lung injury. Am J Respir Crit Care Med. 2006 Jul 15;174(2):187-97. doi: 10.1164/rccm.200506-899OC. Epub 2006 Apr 27. PMID 16645177
- [Background] Mutoh T, Guest RJ, Lamm WJ, Albert RK. Prone position alters the effect of volume overload on regional pleural pressures and improves hypoxemia in pigs in vivo. Am Rev Respir Dis. 1992 Aug;146(2):300-6. doi: 10.1164/ajrccm/146.2.300. PMID 1489116
- [Background] Roldan R, Rodriguez S, Barriga F, Tucci M, Victor M, Alcala G, Villamonte R, Suarez-Sipmann F, Amato M, Brochard L, Tusman G. Sequential lateral positioning as a new lung recruitment maneuver: an exploratory study in early mechanically ventilated Covid-19 ARDS patients. Ann Intensive Care. 2022 Feb 12;12(1):13. doi: 10.1186/s13613-022-00988-9. PMID 35150355
- [Background] Richard JC, Maggiore SM, Mancebo J, Lemaire F, Jonson B, Brochard L. Effects of vertical positioning on gas exchange and lung volumes in acute respiratory distress syndrome. Intensive Care Med. 2006 Oct;32(10):1623-6. doi: 10.1007/s00134-006-0299-y. Epub 2006 Aug 1. PMID 16896856
- [Background] Dellamonica J, Lerolle N, Sargentini C, Hubert S, Beduneau G, Di Marco F, Mercat A, Diehl JL, Richard JC, Bernardin G, Brochard L. Effect of different seated positions on lung volume and oxygenation in acute respiratory distress syndrome. Intensive Care Med. 2013 Jun;39(6):1121-7. doi: 10.1007/s00134-013-2827-x. Epub 2013 Jan 24. PMID 23344832
- [Background] Marrazzo F, Spina S, Forlini C, Guarnieri M, Giudici R, Bassi G, Bastia L, Bottiroli M, Fumagalli R, Langer T. Effects of Trunk Inclination on Respiratory Mechanics in Patients with COVID-19-associated Acute Respiratory Distress Syndrome: Let's Always Report the Angle! Am J Respir Crit Care Med. 2022 Mar 1;205(5):582-584. doi: 10.1164/rccm.202110-2360LE. No abstract available. PMID 34982652
- [Background] Mahran GSK, Abd-Elshafy SK, Abd El Neem MM, Sayed JA. The effect of reference position versus right lateral position on the intra-abdominal pressure in mechanically ventilated patients. Journal of Nursing Education and Practice. 2018;8(6).
- [Background] Vasquez DG, Berg-Copas GM, Wetta-Hall R. Influence of semi-recumbent position on intra-abdominal pressure as measured by bladder pressure. J Surg Res. 2007 May 15;139(2):280-5. doi: 10.1016/j.jss.2006.10.023. Epub 2006 Dec 8. PMID 17161433
- [Background] McBeth PB, Zygun DA, Widder S, Cheatham M, Zengerink I, Glowa J, Kirkpatrick AW. Effect of patient positioning on intra-abdominal pressure monitoring. Am J Surg. 2007 May;193(5):644-7; discussion 647. doi: 10.1016/j.amjsurg.2007.01.013. PMID 17434374
- [Background] Samimian S, Ashrafi S, Khaleghdoost Mohammadi T, Yeganeh MR, Ashraf A, Hakimi H, Dehghani M. The Correlation between Head of Bed Angle and Intra-Abdominal Pressure of Intubated Patients; a Pre-Post Clinical Trial. Arch Acad Emerg Med. 2021 Mar 6;9(1):e23. doi: 10.22037/aaem.v9i1.1065. eCollection 2021. PMID 33870210
- [Background] Selickman J, Crooke PS, Tawfik P, Dries DJ, Gattinoni L, Marini JJ. Paradoxical Positioning: Does "Head Up" Always Improve Mechanics and Lung Protection? Crit Care Med. 2022 Nov 1;50(11):1599-1606. doi: 10.1097/CCM.0000000000005631. Epub 2022 Jul 21. PMID 35866650
- [Background] Wang L, Li X, Yang Z, Tang X, Yuan Q, Deng L, Sun X. Semi-recumbent position versus supine position for the prevention of ventilator-associated pneumonia in adults requiring mechanical ventilation. Cochrane Database Syst Rev. 2016 Jan 8;2016(1):CD009946. doi: 10.1002/14651858.CD009946.pub2. PMID 26743945
- [Background] Guner CK, Kutluturkan S. Role of head-of-bed elevation in preventing ventilator-associated pneumonia bed elevation and pneumonia. Nurs Crit Care. 2022 Sep;27(5):635-645. doi: 10.1111/nicc.12633. Epub 2021 Apr 21. PMID 33884691
- [Background] Marfil-Gomez RM, Garcia-Mayor S, Morales-Asencio JM, Gomez-Gonzalez AJ, Morilla-Herrera JC, Moya-Suarez AB, Aranda-Gallardo M, Rincon-Lopez T, Lupianez-Perez I. Pressure levels in the trochanter area according to repositioning at different degrees of inclination in healthy subjects. J Tissue Viability. 2020 May;29(2):125-129. doi: 10.1016/j.jtv.2020.02.003. Epub 2020 Feb 13. PMID 32115351